CLINICAL TRIAL: NCT04202198
Title: Comparative Evaluation of Recession Coverage Obtained Using Pinhole Surgical Technique, With and With Out Platelet Rich Fibrin : A Randomized Controlled Clinical Trial
Brief Title: Pinhole Surgical Technique for Root Coverage Using PRF
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02_D012_91559
Record Dates: First submitted 2019-12-14; First posted 2019-12-17 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Recession, Gingival
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pinhole surgical technique with Platelet Rich Fibrin (Experimental): minimally invasive tunneling procedure followed by coronal advancement with placement of Platelet Rich Fibrin membrane
  Interventions: Biological: A-PRF
- pinhole surgical technique only (Active Comparator): coronal advancement following minimally invasive tunneling procedure
  Interventions: Procedure: pinhole surgical technique only

INTERVENTIONS:
Biological: A-PRF — local anesthesia was administered followed by placement of a hole in the alveolar mucosa adjacent to mesial most recession tooth. tunneling instruments are used to elevate a full thickness tunnel upto the CEJ sparing the tip of the papilla.previously prepared PRF membranes are placed through the access hole and the flap is advanced. 5-0 polyglycolic acid sutures is used to secure the advanced flap.
  Arms: pinhole surgical technique with Platelet Rich Fibrin
Procedure: pinhole surgical technique only — local anesthesia was administered followed by placement of a hole in the alveolar mucosa adjacent to mesial most recession tooth. tunneling instruments are used to elevate a full thickness tunnel upto the CEJ sparing the tip of the papilla followed by advancement of the flap. 5-0 polyglycolic acid sutures is used to secure the advanced flap.
  Arms: pinhole surgical technique only

SUMMARY:
The current study is a prospective randomised split mouth study to evaluate the effect of Platelet Rich Fibrin as an adjunct to the minimally invasive pinhole surgical technique.

DETAILED DESCRIPTION:
Gingival recession is defined as denudation of the tooth root surface due to the apical movement of the gingiva. The occurrence of gingival recession as a periodontal finding has been estimated to be 78.6%. It is multi-factorial and poses problems from different aspects to the patient.Various etiological factors documented over the years include, (in the decreasing order of frequency) toothbrush trauma, malalignment, local factors, occlusal trauma, high frenum attachment, cervical fillings and crown impingement. Recession levels are also influenced by various other factors such as age, sex, teeth and surfaces of teeth, etc.

Over the years, several authors have presented their views on the etiology, types, treatment modalities and prognosis of gingival recession ranging from the direct lateral sliding flap to the most recent minimally invasive techniques. The1970s saw Harvey and Bernimoulin individually demonstrated the use of coronal advancement of the flap along with the use of grafts with the coronal advancement performed 2 months after the grafting was done on the denuded root surface. Subsequently, over the next 3 decades connective tissue grafts along with coronally advanced flap was established as the gold standard for recession coverage.

Lien-Hui Huang (2005) pioneered the use of blood derivatives in the form of Platelet rich Plasma (PRP) for root coverage but with limited or no substantial improvement over existing techniques. More studies were done on blood derivatives and their efficacy which led to the introduction of the second generation of platelet concentrates, Platelet rich Fibrin, as an alternative. Platelet rich Fibrin was first developed by Choukroun in the year 2001 and has been followed by several studies which have revealed that the slow and sustained release of key growth factors makes it a useful bio-healing material. Comparisons with platelet rich plasma have also proved that, platelet rich fibrin has a better release of growth factors and the presence of leukocytes, which offers quicker and more efficient healing with better regenerative potential.

The recent years have seen newer techniques which are aimed at making it a minimally invasive procedure. One such technique was the pinhole surgical technique given by Chao in the year 2012 which involved a tunnelling procedure along with the usage of a bioresorbable membrane which satisfied the expectations of the trial.6Better outcomes can be achieved with the use patient's own products instead of a foreign graft material. Therefore, the present study compares the effectiveness of Platelet Rich Fibrin as an adjunct to the surgical technique for root coverage

ELIGIBILITY:
Inclusion Criteria:

* Two or more teeth having Millers class I, II andIII or combined recession defects.
* Patients with esthetic concerns and willing to participate in the study
* Age between 18-55 years
* Full mouth plaque score < 20%

Exclusion Criteria:

* Pregnant or lactating females
* Tobacco smokers
* Uncontrolled medical conditions precluding elective surgery
* Untreated periodontal conditions
* Patients treated with any medication known to cause gingival hyperplasia
* Drug and alcohol abuse
* Teeth with hopeless prognosis

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-11-22 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-11-10 (Estimated)

PRIMARY OUTCOMES:
Recession depth reduction | 6 months
  measured as the distance in mm from the CEJ to the gingival margin.
total soft tissue gain | 6 months
  5. Total soft tissue gain (TSTG), measured as the product of gingival recession depth and gingival recession width.
  measured as the product of gingival recession depth and gingival recession width in square mm

SECONDARY OUTCOMES:
mean root coverage | 6 months
  amount of coverage obtained, in percentage

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Rashmi P, MDS, Principal Investigator — Krishnadevaraya college of dental sciences
Locations (1):
- Krishnadevaraya college of dental sciences, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No